CLINICAL TRIAL: NCT07330817
Title: ULTRAVIOLET FIM_A First-In-Man Single Arm Prospective Single Center Study to Assess Safety and Efficacy of Ultra High Pressure PTA Balloon ULTRAVIOLET in Treating A-V Fistula Stenosis
Brief Title: A First-In-Man Study to Assess Safety and Efficacy of Ultra High Pressure PTA Balloon ULTRAVIOLET in Treating A-V Fistula Stenosis
Acronym: ULTRAVIOLETFIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardionovum GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-PER-001
Record Dates: First submitted 2025-12-11; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Arterio-venous Fistula; Stenosis of Arteriovenous Dialysis Fistula
Keywords: A-V fistula; First-In-Man; Ultra-High Pressure Balloon; PTA balloon; Resistant Stenotic Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ULTRAVIOLET UHP PTA (Experimental): Percutaneous transluminal angioplasty with ultra-high-pressure balloon
  Interventions: Device: PTA balloon

INTERVENTIONS:
Device: PTA balloon — Angioplasty of a resistant stenotic lesion in the arterio-venous fistula

SUMMARY:
First-In-Man Single Arm Prospective Study to assess the safety and efficacy of ULTRAVIOLET UHP PTA balloon.

DETAILED DESCRIPTION:
First-In-Man Single Site study to assess safety and efficacy of ultra-high pressure PTA balloon called ULTRAVIOLET UHP PTA in treating resistant stenotic lesions in arterio-venous fistula of dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand the purpose of the study, voluntarily agree to participate and signed Informed Consent form
* Patients with impaired haemodialysis access due to narrowed lesions, as indicated by contrast or ultrasound or clinical diagnosis.
* Indications for percutaneous endovascular therapy with diameter stenosis >50% and fistula's hemodynamic showing abnormalities (thrombosis in the AVF, high venous pressure, re-circulation, abnormal physical examination, decrease in dialysis efficiency, decrease in blood flow through the vascular access)
* Target lesion is a resistant de novo or restenotic lesion
* The target lesion is located in the reflux vein from the anastomotic site of arteriovenous fistula (AVF) to the distal end of the subclavian vein (excluding the anastomotic site of AVF); if there are no target lesions, they should be treated with standard angioplasty balloon before treating the target lesion.

Exclusion Criteria:

* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrolment into this study;
* Patients who are actively participating in another drug or device investigational study, who have not completed the primary endpoint follow-up period;
* Patients who have undergone major surgical procedures (such as open chest surgery, head surgery) within 30 days before being enrolled in the study;
* Patients who plan to undergo major surgical procedures (such as open chest surgery, head surgery) within 30 days after being enrolled in the study;
* Immature AVF (not used for dialysis; due to insufficient inner diameter, inability to ensure successful puncture, and inadequate blood flow, this access has not been used for successful dialysis);
* AVF has been implanted with a stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Technical Success | At the end of the procedure (up to 40 minutes)
  Ability to cross the lesion and fully efface the balloon, leaving no residual stenosis (<30%) evaluated by fistulography
Freedom from procedure-related complications after 1 month | 1 month
  freedom from adverse events related to the procedure in 1 month follow up period

SECONDARY OUTCOMES:
Acute Device Success | At the end of the procedure (up to 40 minutes)
  successful delivery, balloon inflation, deflation, and retrieval of the intact study device without burst below rated burst pressure
Clinical Success | At the end of the procedure (up to 40 minutes)
  after intervention, the function of hemodialysis access is improved, dialysis function is restored, and at least one complete dialysis session has been completed
Procedural Surgery success | At the end of hospitalization (assessed up to 5 days)
  Once technical success has been achieved, no major adverse events (MAE) occurred during the procedure or hospitalization, including death, stroke, thrombosis, allergic reactions, or pulmonary disease
Target Lesion Primary Patency | 1 month
  Primary patency rate refers to the peak systolic velocity ratio (PSVR) measured by Doppler ultrasound (DUS) ≤ 2.0, which confirms the absence of restenosis and does not require clinically driven target lesion revascularization (CD-TLR)
Freedom from target lesion revascularization | 1 month
  Clinical symptoms and dialysis indicators indicate that dialysis cannot be successfully performed, and the target lesion location (confirmed by Doppler ultrasound) +/-5 mm proximal/distal requires re-intervention surgery
Major Adverse Events (MAE) | 1 month
  Occurrence of major adverse events (MAE)
Dialysis Circuit Patency | 1 month
  Patency of the whole patency circuit evaluated at Doppler Ultra-Sound (DUS)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Tozzi, MD, PhD, Principal Investigator — Universita' Insubria, ASST Sette Laghi, Varese, Italy
Locations (1):
- ASST Sette Laghi, Varese, Italy

IPD SHARING:
Plan to Share IPD: No